CLINICAL TRIAL: NCT03153943
Title: HIP Mobile: A Community-based Monitoring, Rehabilitation and Learning e-System for Patients Following a Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Greybox Solutions Inc. (Unknown)
Responsible Party: Principal Investigator, Suzanne Morin, Dr., McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-248-MUHC
Record Dates: First submitted 2017-05-10; First posted 2017-05-15 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workbook support group (Experimental): Printed educational workbook and pedometer.
  Interventions: Other: Workbook support
- HIP Mobile e-Monitoring support group (Experimental): Remote monitoring via smart shoe insoles and a coaching with enabling educational electronic program accessed through a tablet.
  Interventions: Device: HIP Mobile e-Monitoring support

INTERVENTIONS:
Device: HIP Mobile e-Monitoring support — 3-month community-based extended-rehabilitation e-Monitoring and Coaching support program
  Arms: HIP Mobile e-Monitoring support group
Other: Workbook support — Printed material support
  Arms: Workbook support group

SUMMARY:
Approximately 30,000 adults in Quebec over the age of 50 suffer a fragility fracture each year. Fractures can affect a person's health, well-being and autonomy. Personal costs of these fractures are high, with as many as 50% of hip fracture patients being unable to return their pre-fracture level of autonomy.

Homecare and community services provide customary rehabilitation support immediately following discharge from acute-care, though this contribution can be limited by lack of resources. For those patients at risk of negative outcomes, we have demonstrated clinically important benefits of extended exercise rehabilitation programs offered beyond the regular rehabilitation period on improving physical function.

Through advances in sensor and telecommunication technology, eHealth solutions incorporated within homecare services as an integral part of the continuum of care can lead to better patient and health professional experience, improve clinical outcomes and reduce costs to the healthcare system.

The purpose of this study is to determine if the implementation of a 3-month community-based extended-rehabilitation e-Monitoring and Coaching support program is more effective at improving mobility in community-dwelling elderly patients who have sustained a fracture than a printed material support program, and if these effects persist 6 months after discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling men and women aged ≥ 60 years
* Treated for any fracture excluding hands, feet, patella, cervical spine, skull, ribs, or clavicle, at any of the 3 participating sites, within the previous 8 weeks.

Exclusion Criteria:

* Upper limb fractures that do not meet the criteria of gait frailty
* Multiple traumas
* Open fractures
* Pathological fractures
* Inability to communicate adequately in either French or English
* Inability to give written informed consent
* Discharge to a long-term care institution

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Change in mobility | 0, 1, 3, and 7 months
  Measured as an ordinal mobility response variable quantified by the number of minimal clinically important changes (MIC) a participant attains using the gait speed and 30 second Sit to Stand tests. A person making no MIC in either measure is given a response category of 0, the lowest. A person changing by 1 MIC on only of the measures (either one) will be given a value of 1; a MIC gain on both measures would be assigned a value of 2, and so forth.

SECONDARY OUTCOMES:
Change in grip strength | 0, 1, 3, and 7 months
  Measured using a Jamar™ hand dynamometer.
Change in walking endurance | 0, 1, 3, and 7 months
  Measured using the 2-minute walk test.
Change in balance | 0, 1, 3, and 7 months
  Measured using the Berg Balance Scale.
Change in the spatial area an individual moves through | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 months
  Measured using the Life Space Mobility Assessment
Change in global function status | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 months
  Measured using the Reintegration to Normal Living Index (RNLI)
Change in perceived physical health status | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 months
  Measured by the physical function subscale of the RAND-36
Change in Health-related quality of life | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 months
  Measured by the EQ-5D
Change in patient-reported health perception | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 months
  Measured by the How Are You Today? Visual Analog Health States
Change in goal directed behavior | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 months
  Measured by the Apathy Evaluation Scale
Change in global quality of life (QOL) | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 months
  Measured by Patient Generated Index (PGI)
Change in cognition | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 months
  Measured by the Perceived Deficits Questionnaire (PDQ)
Change in confidence in maintaining balance while doing daily activities. | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 months
  Measured by the Activities-specific Balance Confidence Scale (ABC-S)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Morin, MD, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (3):
- Canada (3):
  - McGill University Health Centre, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No